CLINICAL TRIAL: NCT01720576
Title: Study to Assess the Safety and Tolerability of Multiple Ascending Doses of REGN1033 (SAR391786)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1033-HV-1204
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Dose 1 of REGN1033 (SAR391786) or Placebo
  Interventions: Drug: REGN1033 (SAR391786); Drug: Placebo
- Cohort 2 (Experimental): Dose 2 of REGN1033 (SAR391786) or Placebo
  Interventions: Drug: REGN1033 (SAR391786); Drug: Placebo
- Cohort 3 (Experimental): Dose 3 of REGN1033 (SAR391786) or Placebo
  Interventions: Drug: REGN1033 (SAR391786); Drug: Placebo

INTERVENTIONS:
Drug: REGN1033 (SAR391786)
Drug: Placebo

SUMMARY:
This is a study to assess the safety and tolerability of subcutaneously administered REGN1033 (SAR391786) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects are males and females aged 60 years and older with no significant health issues or clinically significant abnormal laboratory values.

A subject must meet the following criteria to be eligible for inclusion in the study:

1. Sexually active males willing to use contraceptives during the study and through 4 months after the study.
2. Female subjects not of child bearing potential (surgically sterile or postmenopausal for longer than 1 year)
3. Body mass index (BMI) between 18.5 and 32 kg/m2 inclusive
4. Willing to maintain current diet and exercise routine for the duration of the study
5. Willing and able to return for all clinic visits and complete all study-related procedures
6. Able to read and understand, and willing to sign the ICF

Exclusion Criteria:

1. Significant concomitant illness such as, but not limited to cardiac, renal, rheumatologic, gastrointestinal, hematological, skeletal/muscular, neurologic, psychiatric, endocrine, metabolic or immunological disease.
2. Evidence of malnutrition
3. Cachexia of any cause
4. Evidence or history of muscle diseases or weakness with the exception of age related muscle loss
5. Limb amputation
6. Immobilization, surgical procedure, fracture, or trauma to the upper or lower limb within 6 months
7. History or evidence of heart diseases including but not limited to coronary heart disease with/without history of myocardial infarction, chronic or acute heart failure (New York Heart Association [NYHA] stage 2-4), cardiac arrhythmia with clinical symptoms, valvular heart disease, and cardiac hypertrophy of clinical significance
8. Women of childbearing potential (not surgically sterile or amenorrheic for at least 12 months if postmenopausal)
9. Uncontrolled diabetes defined as HbA1C > 7.5 at screening; if taking oral hypoglycemic drugs, have to be on stable doses of medication for more than 3 months. Diabetics using insulin are excluded
10. Asthmatic subjects with current or recurring symptoms within 1 year.
11. History of, COPD, chronic kidney disease, cancer except primary basal-cell skin cancer that has been adequately treated
12. Neurological injury (eg, stroke) within 1 year
13. Abnormal or uncontrolled blood pressure at screening visit defined as diastolic BP >95 and/or systolic BP >160 mm Hg; if taking hypertensive medication, have to be on stable doses of medication for more than 3 months
14. Hepatic transaminases (ALT and or AST) > 2X ULN
15. Reduced renal function as defined by eGFR<60 mL/min
16. Current smokers or previous smokers who stopped smoking within 6 months
17. Current or recent history (within 1 year of screen) of alcohol or drug abuse
18. History of hypersensitivity response to any biologics
19. History of hypersensitivity to doxycycline or other tetracycline antibiotics
20. Current or recent participation in any clinical trial (within 30 days of small molecular drugs or within 3 months of biologics)
21. Exposure within 3 months to approved biological drugs. (The name of the drug and duration of previous exposure will be recorded). Vaccines are allowed.
22. Sexually active men* who are unwilling to practice adequate contraception during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs | Day 1 to Day 141
  The primary endpoint in the study is the incidence and severity of TEAEs (Treatment Emergent Adverse Events) in participants treated with REGN1033 (SAR391786) or placebo, reported from the time of administration of study drug on day 1 (baseline) to day 141 (end of study).

SECONDARY OUTCOMES:
Serum concentration of REGN1033 (SAR391786) | Day 1 to Day 141
  Serum concentration of REGN1033 (SAR391786) over time
immunogenicity | Day 1 to Day 141
  Presence or absence of anti-REGN1033 (SAR391786) antibodies over time (immunogenicity )

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Daytona Beach, Florida
  - Evansville, Indiana